CLINICAL TRIAL: NCT04585022
Title: Whole Blood Metal Ion Concentrations in Metal-on-metal Total Hip Arthroplasty and Hip Resurfacing - A Randomized Controlled Trial With 5-years Follow up Including 75 Patients
Brief Title: Whole Blood Metal Ion Concentrations in Metal-on-metal Total Hip Arthroplasty and Hip Resurfacing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High early failure rates and adverse reactions in similar devices
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Anders Troelsen, MD, PhD, dr.med., Professor, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KF 01-309171
Record Dates: First submitted 2020-09-23; First posted 2020-10-14 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Hip
Keywords: Metal ion concentration; Total hip arthroplasty; Hip resurfacing
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both the care provider and patient were blinded until day of surgery. The laboratory analyzing blood metal concentrations were blinded to treatment allocation throughout the study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnum (Active Comparator): A metal-on-metal large diameter head total hip arthroplasty
  Interventions: Device: Magnum, Zimmer Biomet, Warsaw, IN
- Recap (Active Comparator): A metal-on-metal hip resurfacing arthroplasty
  Interventions: Device: Recap, Zimmer Biomet, Warsaw, IN

INTERVENTIONS:
Device: Magnum, Zimmer Biomet, Warsaw, IN
  Arms: Magnum
Device: Recap, Zimmer Biomet, Warsaw, IN
  Arms: Recap

SUMMARY:
The investigators aimed to investigate the possible differences in metal ion concentrations in patients following one of two types of metal-on-metal articulating hip prosthesis regarding chromium and cobalt concentration, radiological findings, patient reported outcome measures and rate of revision at 5-years follow up.

DETAILED DESCRIPTION:
The metal-on-metal large-diameter-head (MoM-LDH) hip replacements increased in popularity during the start of the 21st century. Subsequently reports raised concerns regarding adverse reactions due to elevated chromium (Cr) and cobalt (Co) concentrations as well as high rates of other complications and revisions.

This was a single center parallel-group randomized controlled trial. The primary outcome was to compare Cr and Co concentrations at 5-years follow up following MoM-LDH total hip arthroplasty (MoM-LDH-THA) or MoM-LDH hip resurfacing (MoM-LDH-HR).

Secondary outcomes were radiological findings, patient reported outcome measures and revision rate at 5-years follow up.

The study was prematurely terminated in 2012 due to alerts and safety communications from the Danish national regulatory agency regarding early failure rates and high incidence of ARMD in patients with MoM hip implants [13]. At that time the study population consisted of 75 patients out of 200 planned for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary hip osteoarthritis eligible for hip replacement surgery
* Able to give informed consent
* Able to complete follow up consultations

Exclusion Criteria:

* Earlier or present infection of the hip
* Severe systemic or metabolic disease leading to weakening of the bone
* Severe congenital hip dysplasia
* Osteoporosis and/or renal disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, MD, Principal Investigator — Hvidovre University Hospital

IPD SHARING:
Plan to Share IPD: No
No IPD are to be shared with other researchers.

REFERENCES:
- [Background] Schmalzried TP, Peters PC, Maurer BT, Bragdon CR, Harris WH. Long-duration metal-on-metal total hip arthroplasties with low wear of the articulating surfaces. J Arthroplasty. 1996 Apr;11(3):322-31. doi: 10.1016/s0883-5403(96)80085-4. PMID 8713913
- [Background] Chan FW, Bobyn JD, Medley JB, Krygier JJ, Tanzer M. The Otto Aufranc Award. Wear and lubrication of metal-on-metal hip implants. Clin Orthop Relat Res. 1999 Dec;(369):10-24. doi: 10.1097/00003086-199912000-00003. PMID 10611857
- [Background] Cuckler JM, Moore KD, Lombardi AV Jr, McPherson E, Emerson R. Large versus small femoral heads in metal-on-metal total hip arthroplasty. J Arthroplasty. 2004 Dec;19(8 Suppl 3):41-4. doi: 10.1016/j.arth.2004.09.006. PMID 15578551
- [Background] Peters CL, McPherson E, Jackson JD, Erickson JA. Reduction in early dislocation rate with large-diameter femoral heads in primary total hip arthroplasty. J Arthroplasty. 2007 Sep;22(6 Suppl 2):140-4. doi: 10.1016/j.arth.2007.04.019. Epub 2007 Jul 27. PMID 17823033
- [Background] Papageorgiou I, Yin Z, Ladon D, Baird D, Lewis AC, Sood A, Newson R, Learmonth ID, Case CP. Genotoxic effects of particles of surgical cobalt chrome alloy on human cells of different age in vitro. Mutat Res. 2007 Jun 1;619(1-2):45-58. doi: 10.1016/j.mrfmmm.2007.01.008. Epub 2007 Jan 25. PMID 17376492
- [Background] Langton DJ, Joyce TJ, Jameson SS, Lord J, Van Orsouw M, Holland JP, Nargol AV, De Smet KA. Adverse reaction to metal debris following hip resurfacing: the influence of component type, orientation and volumetric wear. J Bone Joint Surg Br. 2011 Feb;93(2):164-71. doi: 10.1302/0301-620X.93B2.25099. PMID 21282753
- [Background] Whitehouse MR, Aquilina AL, Patel S, Eastaugh-Waring SJ, Blom AW. Survivorship, patient reported outcome and satisfaction following resurfacing and total hip arthroplasty. J Arthroplasty. 2013 May;28(5):842-8. doi: 10.1016/j.arth.2013.01.007. Epub 2013 Mar 13. PMID 23489727
- [Background] Langton DJ, Jameson SS, Joyce TJ, Hallab NJ, Natu S, Nargol AV. Early failure of metal-on-metal bearings in hip resurfacing and large-diameter total hip replacement: A consequence of excess wear. J Bone Joint Surg Br. 2010 Jan;92(1):38-46. doi: 10.1302/0301-620X.92B1.22770. PMID 20044676
- [Background] Bozic KJ, Kurtz S, Lau E, Ong K, Chiu V, Vail TP, Rubash HE, Berry DJ. The epidemiology of bearing surface usage in total hip arthroplasty in the United States. J Bone Joint Surg Am. 2009 Jul;91(7):1614-20. doi: 10.2106/JBJS.H.01220. PMID 19571083
- [Background] Mahomed NN, Arndt DC, McGrory BJ, Harris WH. The Harris hip score: comparison of patient self-report with surgeon assessment. J Arthroplasty. 2001 Aug;16(5):575-80. doi: 10.1054/arth.2001.23716. PMID 11503116
- [Background] DeLee JG, Charnley J. Radiological demarcation of cemented sockets in total hip replacement. Clin Orthop Relat Res. 1976 Nov-Dec;(121):20-32. PMID 991504
- [Background] Gruen TA, McNeice GM, Amstutz HC. "Modes of failure" of cemented stem-type femoral components: a radiographic analysis of loosening. Clin Orthop Relat Res. 1979 Jun;(141):17-27. PMID 477100
- [Background] Callanan MC, Jarrett B, Bragdon CR, Zurakowski D, Rubash HE, Freiberg AA, Malchau H. The John Charnley Award: risk factors for cup malpositioning: quality improvement through a joint registry at a tertiary hospital. Clin Orthop Relat Res. 2011 Feb;469(2):319-29. doi: 10.1007/s11999-010-1487-1. PMID 20717858
- [Background] Borgwardt A, Borgwardt L, Zerahn B, Daugaard H, Borgwardt L, Ribel-Madsen S. A Randomized Seven-Year Study on Performance of the Stemmed Metal M2a-Magnum and Ceramic C2a-Taper, and the Resurfacing ReCap Hip Implants. J Arthroplasty. 2018 May;33(5):1412-1420. doi: 10.1016/j.arth.2017.11.061. Epub 2017 Dec 5. PMID 29276121
- [Background] Costa ML, Achten J, Parsons NR, Edlin RP, Foguet P, Prakash U, Griffin DR; Young Adult Hip Arthroplasty Team. Total hip arthroplasty versus resurfacing arthroplasty in the treatment of patients with arthritis of the hip joint: single centre, parallel group, assessor blinded, randomised controlled trial. BMJ. 2012 Apr 19;344:e2147. doi: 10.1136/bmj.e2147. PMID 22517930
- [Background] Garbuz DS, Tanzer M, Greidanus NV, Masri BA, Duncan CP. The John Charnley Award: Metal-on-metal hip resurfacing versus large-diameter head metal-on-metal total hip arthroplasty: a randomized clinical trial. Clin Orthop Relat Res. 2010 Feb;468(2):318-25. doi: 10.1007/s11999-009-1029-x. Epub 2009 Aug 21. PMID 19697090
- [Background] Khan M, Kuiper JH, Sieniawska C, Richardson JB. Differences in concentration of metal debris in blood, serum, and plasma samples of patients with metal-on-metal hip resurfacing arthroplasty. J Orthop. 2015 Dec 9;13(4):450-454. doi: 10.1016/j.jor.2015.10.006. eCollection 2016 Dec. PMID 27857480
- [Background] Jantzen C, Jorgensen HL, Duus BR, Sporring SL, Lauritzen JB. Chromium and cobalt ion concentrations in blood and serum following various types of metal-on-metal hip arthroplasties: a literature overview. Acta Orthop. 2013 Jun;84(3):229-36. doi: 10.3109/17453674.2013.792034. Epub 2013 Apr 18. PMID 23594249
- [Background] Renner L, Faschingbauer M, Schmidt-Braekling T, Boettner F. Cobalt serum levels differ in well functioning Birmingham resurfacing and Birmingham modular THA. Arch Orthop Trauma Surg. 2016 May;136(5):715-21. doi: 10.1007/s00402-016-2439-3. Epub 2016 Mar 16. PMID 26983720
- [Background] Hutt J, Lavigne M, Lungu E, Belzile E, Morin F, Vendittoli PA. Comparison of Whole-Blood Metal Ion Levels Among Four Types of Large-Head, Metal-on-Metal Total Hip Arthroplasty Implants: A Concise Follow-up, at Five Years, of a Previous Report. J Bone Joint Surg Am. 2016 Feb 17;98(4):257-66. doi: 10.2106/JBJS.O.00201. PMID 26888673
- [Background] Jacobs JJ, Skipor AK, Patterson LM, Hallab NJ, Paprosky WG, Black J, Galante JO. Metal release in patients who have had a primary total hip arthroplasty. A prospective, controlled, longitudinal study. J Bone Joint Surg Am. 1998 Oct;80(10):1447-58. doi: 10.2106/00004623-199810000-00006. PMID 9801213
- [Background] Berstock JR, Whitehouse MR, Duncan CP. Trunnion corrosion: what surgeons need to know in 2018. Bone Joint J. 2018 Jan;100-B(1 Supple A):44-49. doi: 10.1302/0301-620X.100B1.BJJ-2017-0569.R1. PMID 29292339
- [Background] Varnum C, Pedersen AB, Makela K, Eskelinen A, Havelin LI, Furnes O, Karrholm J, Garellick G, Overgaard S. Increased risk of revision of cementless stemmed total hip arthroplasty with metal-on-metal bearings. Acta Orthop. 2015;86(4):469-76. doi: 10.3109/17453674.2015.1023132. Epub 2015 Feb 26. PMID 25715878
- [Background] Junnila M, Kostensalo I, Virolainen P, Remes V, Matilainen M, Vahlberg T, Pulkkinen P, Eskelinen A, Itala A, Makela K. Hip resurfacing arthroplasty versus large-diameter head metal-on-metal total hip arthroplasty: comparison of three designs from the Finnish Arthroplasty Register. Scand J Surg. 2014 Mar;103(1):54-9. doi: 10.1177/1457496913495345. Epub 2013 Dec 17. PMID 24345980
- [Background] Jack CM, Walter WL, Shimmin AJ, Cashman K, de Steiger RN. Large diameter metal on metal articulations. Comparison of total hip arthroplasty and hip resurfacing arthroplasty. J Arthroplasty. 2013 Apr;28(4):650-3. doi: 10.1016/j.arth.2012.07.032. Epub 2012 Nov 7. PMID 23140992
- [Derived] Hersnaes PN, Gromov K, Otte KS, Gebuhr PH, Troelsen A. Harris Hip Score and SF-36 following metal-on-metal total hip arthroplasty and hip resurfacing - a randomized controlled trial with 5-years follow up including 75 patients. BMC Musculoskelet Disord. 2021 Sep 12;22(1):781. doi: 10.1186/s12891-021-04671-1. PMID 34511090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a tertiary health care center in Copenhagen, Denmark from November 2006 to January 2012. 5-years follow up consultations were conducted from 2011 to 2017.
Groups:
- Magnum: A metal-on-metal large diameter head total hip arthroplasty
  Magnum, Zimmer Biomet, Warsaw, IN
- Recap: A metal-on-metal hip resurfacing arthroplasty
  Recap, Zimmer Biomet, Warsaw, IN
Period: Overall Study
Arm/Group | Magnum | Recap
Started | 39 | 36
Completed | 33 | 25
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnum | Recap | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.9 [56.5 to 63.2] | 59.4 [51.2 to 63.58] | 60.8 [54.55 to 63.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 26 | 26 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 39 | 36 | 75
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 28.4 [25.8 to 28.93] | 27.45 [24.6 to 29.32] | 27.9 [25.2 to 31.0]

OUTCOME MEASURES:

1. Primary Outcome: Metal Ion Concentrations in Blood
Description: Chromium and cobalt concentrations in whole blood
Time Frame: at 5 years follow up
Population: The discrepancy between numbers of patients analysed and the numbers presented in Participant flow is due to patients who had bilateral MoM hip replacement at the 5-year follow-up were excluded in addition to those lost to follow up, who had revision surgery or died before 5-years follow up.
Measure: Median (Inter-Quartile Range); unit: micrograms/liter
Arm/Group | Magnum | Recap
Number analyzed (Participants) | 25 | 20
micrograms/liter
  Chromium | 1.36 [0.99 to 3.11] | 1.21 [0.88 to 3.03]
  Cobalt | 1.67 [0.86 to 2.31] | 0.92 [0.64 to 1.49]

2. Secondary Outcome: Harris Hip Score
Description: Harris Hip Score (0-100, higher values meaning better outcome)
Time Frame: at 5 years follow up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Magnum | Recap
Number analyzed (Participants) | 33 | 25
units on a scale | 100 [98 to 100] | 100 [93 to 100]

3. Secondary Outcome: SF-36
Description: Short Form 36 Health Survey Questionnaire (SF-36) (0-100, higher values meaning better outcome)
Time Frame: at 5 years follow up
Population: The total number of patients analyzed is different from the total number of patients who completed the study, since some patients had missing data for this questionnaire.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Magnum | Recap
Number analyzed (Participants) | 30 | 26
score on a scale
  Physical function | 90 [68.75 to 95] | 90 [70 to 100]
  Physical restriction | 100 [66.67 to 100] | 100 [50 to 100]
  Bodily pain | 92 [62 to 100] | 84 [62 to 100]
  General health | 74.5 [61.75 to 89.25] | 79.5 [56.44 to 87]
  Vitality | 77.5 [60 to 85] | 75 [32.5 to 85]
  Social function | 100 [100 to 100] | 100 [100 to 100]
  Emotional restriction | 100 [100 to 100] | 100 [100 to 100]
  Mental Health | 92 [72 to 96] | 88 [76 to 92]

4. Secondary Outcome: Number of Patients Undergoing Revision
Description: Rate of revision during the follow-up period, calculated as number of revisions (numerator) out of the total number of patients starting the study (denominator)
Time Frame: at 5 years follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Magnum | Recap
Number analyzed (Participants) | 39 | 36
Participants | 0 | 6

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Magnum | Recap
All-Cause Mortality (participants affected / at risk) | 2/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/39 | 6/36
Other Adverse Events (participants affected / at risk) | 0/39 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnum (N=39) | Recap (N=36)
Septic loosening of stem (Infections and infestations) | 0 (0) | 1 (1)
Fracture of femoral neck (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Unexplained hip pain without joint failure (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aseptic loosening of cup (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
adverse reaction to metal debris (Product Issues) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to a revision rate of 16.7% in the MoM-HR group and lost at follow up (15.4% and 13.9% for MoM-LDH-THA and MoM-HR respectively) in both groups data were not complete.

No preoperative data were obtained for our primary or secondary outcomes. Due to premature termination of the study it lacks power causing a risk of type II error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No